CLINICAL TRIAL: NCT04094766
Title: A Phase I Clinical Study of Dual Specificity CD19 and CD22 Chimeric Antigen Receptor T Cell Therapy in Relapsed or Refractory Acute B Lymphoblastic Leukemia
Brief Title: Safety and Efficacy of Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy in R/R Acute B Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Production plan adjustment
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU-BLLCAR-L10D
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Refractory B Acute Lymphoblastic Leukemia; Relapse B Acute Lymphoblastic Leukemia
Keywords: Chimeric Antigen Receptor T cells; CD19 and CD22
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BLLCAR-L10D treatment group (Experimental): In BLLCAR-L10D treatment group, patients will be treated with dual specificity CD19 and CD22 CAR-T cells with a escalation approach, 3 CAR-T dosage will be tested in this study: 0.5×10^6, 1.5×10^6, 2.0×10^6 CAR-T cells/kg.
  Interventions: Drug: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy

INTERVENTIONS:
Drug: Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy — Patients will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of CAR-T cells. After a pre-treatment lymphodepletion therapy, patients will receive the Dual Specificity CD19 and CD22 CAR-T Cell Immunotherapy by intravenous injection.

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and efficacy of infusion of dual specificity CD19 and CD22 CAR-T cells in patients with relapsed and refractory acute B lymphoblastic leukemia.

DETAILED DESCRIPTION:
CD19-directed CAR-T cell therapy has shown promising results for the treatment of relapsed or refractory acute B lymphoblastic leukemia. CD19 and CD22 are proteins usually expressed on the surface of the B leukemia cells. The dual specificity CAR enables the T-cells to recognize and kill the tumor cell through recognition of CD19 and CD22.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent could be acquired;
2. Diagnosed with relapse/refractory acute lymphoblastic leukemia;
3. Relapse was defined as recurrence of blast cell(more than 5%) in peripheral blood or in bone marrow or extramedullary involvement;
4. Refractory was defined as failed to achieve complete remission after two courses of induction therapy;
5. CD19/CD22 postive leukemia cell was confirmed by flow cytometry or immunohistochemistry within 90 days since enrollment in this trial;
6. Karnofsky score ≥70;
7. Results of pregnant test should be negative, and agree to conception control during treatment and 6 months after CAR-T infusion.
8. Adequate organ function: EF≥50%; normal ECG; CCR ≥ 50ml/min or Cr < 2.0mg/dL or < 2 times upper limitation of normal; ALT and AST<5 times upper limitation of normal; Serum bilirubin ≤ 3.0mg/dL; DLCO or FEV1 > 45% of predict value;
9. At least 2 weeks intervals since the last chemotherapy;
10. At least 2 weeks intervals since the last anti-GVHD therapy if patients have ever ;

Exclusion Criteria:

1. Patients diagnosed with acute promyelocytic leukemia:t(15;17)(q22;q12);
2. Women in pregnancy and lactation;
3. Uncontrolled infection, Active HBV or HCV infection, HIV positive or any other deadly bacterial/virual diseases;
4. Long term use of systemic corticosteroids(5mg per day for 2 weeks);
5. Any other uncontrolled life-threaten diseases;
6. Patients with history of anaphylaxis to any drugs;
7. With central nervous system (CNS) involvement;
8. Patients with GVHD after allo-HSCT who needed immunosuppressive agents ;
9. Patients with acute autoimmune diseases such as psoriasis or rheumatoid arthritis;
10. Other conditions that principle investigator considered may increase the risk of the patients or interference the results.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events | Day 1-100 days after injection
  Assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Objective response rate | Day 1-5 years after injection
  Objective response include complete remission and partial remission
Overall survival | Day 1-5 years after injection
Progression free survival | Day 1-5 years after injection

OTHER OUTCOMES:
Copy numbers of CAR-T cells in patients | Day 1-5 years after injection

CONTACTS AND LOCATIONS:
Overall Officials: Aili He, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided